CLINICAL TRIAL: NCT04783064
Title: Association Between Anatomic Characteristics of Neck and Diaphragmatic Palsy After Brachial Plexus Block: A Prospective Observational Study
Brief Title: Neck Anatomy and Phrenic Nerve Palsy After BPB
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: H-2102-133-1199
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Diaphragm; Paralysis
MeSH Terms: conditions — Respiratory Paralysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — Interscalene brachial plexus block is performed at ipsilateral side of the affected shoulder.

SUMMARY:
The purpose of this study was to determine the association between the anatomical characteristics of neck and postoperative diaphragmatic paralysis in patients undergoing interscalene brachial plexus block before shoulder arthroscopic surgery.

DETAILED DESCRIPTION:
The purpose of this study was to determine the association between the anatomical characteristics of neck and postoperative diaphragmatic paralysis in patients undergoing interscalene brachial plexus block before shoulder arthroscopic surgery. In addition, we want to identify risk factors for diaphragmatic paralysis after brachial plexus block. Through this study, we can find the basis for predicting the possibility of diaphragmatic paralysis after brachial plexus block according to the patient's anatomical characteristics and procedural factors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 19 years undergoing shoulder arthroscopic surgery for a rotator cuff tear repair under general anesthesia

Exclusion Criteria:

* Patients who refused to participate in the trial

  * Patients with respiratory diseases such as asthma and chronic obstructive pulmonary disease

    * Patients with neurological abnormalities of the upper limb

      * Patients with a history of surgery around the neck on the ipsilateral side of the surgery site, radiation treatment history, etc.

        * Patients with a history of allergy or hypersensitivity reactions to local anesthetics

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over 19 years undergoing shoulder arthroscopic surgery for a rotator cuff tear repair under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Phrenic nerve palsy | 10 minutes after the end of surgery
  Ultrasound is used to check the movement of the diaphragm on the operation side. The movement of the diaphragm is measured in centimeters when checked with M-mode in a forceful sniffing state.

SECONDARY OUTCOMES:
Neck length | Before induction, 1-2 minutes
  The neck length is measured by drawing a straight line from the mandible angle on the side to the middle point of the clavicle with a tape measure.
Neck girth | Before induction, 1-2 minutes
  The neck circumference length is measured by a tape ruler over the upper plane of the spinous process of the 7th cervical spine at the back and the lower plane of the thyroid cartilage at the front side in the patient's sitting position.
Height | At admission, 1-2 minutes
  Height (cm)
Weight | At admission, 1-2 minutes
  Weight (kg)
Sex | At admission, 1-2 minutes
  Sex
The method of brachial plexus block | During brachial plexus block, 10 minutes
  Specific location where the brachial plexus block was performed (Specific location of needle tip where local anesthetic is injected)
The volume (dose) of local anesthetics injected | During brachial plexus block, 10 minutes
  The volume (dose) of local anesthetics injected

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, M.D, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Kim DH, Lin Y, Beathe JC, Liu J, Oxendine JA, Haskins SC, Ho MC, Wetmore DS, Allen AA, Wilson L, Garnett C, Memtsoudis SG. Superior Trunk Block: A Phrenic-sparing Alternative to the Interscalene Block: A Randomized Controlled Trial. Anesthesiology. 2019 Sep;131(3):521-533. doi: 10.1097/ALN.0000000000002841. PMID 31283740
- [Background] Lee JH, Cho SH, Kim SH, Chae WS, Jin HC, Lee JS, Kim YI. Ropivacaine for ultrasound-guided interscalene block: 5 mL provides similar analgesia but less phrenic nerve paralysis than 10 mL. Can J Anaesth. 2011 Nov;58(11):1001-6. doi: 10.1007/s12630-011-9568-5. Epub 2011 Aug 20. PMID 21858614
- [Background] Kang R, Jeong JS, Chin KJ, Yoo JC, Lee JH, Choi SJ, Gwak MS, Hahm TS, Ko JS. Superior Trunk Block Provides Noninferior Analgesia Compared with Interscalene Brachial Plexus Block in Arthroscopic Shoulder Surgery. Anesthesiology. 2019 Dec;131(6):1316-1326. doi: 10.1097/ALN.0000000000002919. PMID 31490292
- [Background] Bao X, Huang J, Feng H, Qian Y, Wang Y, Zhang Q, Hu H, Wang X. Effect of local anesthetic volume (20 mL vs 30 mL ropivacaine) on electromyography of the diaphragm and pulmonary function after ultrasound-guided supraclavicular brachial plexus block: a randomized controlled trial. Reg Anesth Pain Med. 2019 Jan;44(1):69-75. doi: 10.1136/rapm-2018-000014. PMID 30640655
- [Background] Choi JH, Miyazaki S, Okawa M, Kim EJ, Ryu JJ, Lee JB, Shin C, Lee SH. Clinical implications of mandible and neck measurements in non-obese asian snorers: ansan city general population-based study. Clin Exp Otorhinolaryngol. 2011 Mar;4(1):40-3. doi: 10.3342/ceo.2011.4.1.40. Epub 2011 Mar 17. PMID 21461062
- [Background] Zhang Y, Wu H, Xu Y, Qin H, Lan C, Wang W. The correlation between neck circumference and risk factors in patients with hypertension: What matters. Medicine (Baltimore). 2020 Nov 20;99(47):e22998. doi: 10.1097/MD.0000000000022998. PMID 33217801
- [Background] El-Boghdadly K, Chin KJ, Chan VWS. Phrenic Nerve Palsy and Regional Anesthesia for Shoulder Surgery: Anatomical, Physiologic, and Clinical Considerations. Anesthesiology. 2017 Jul;127(1):173-191. doi: 10.1097/ALN.0000000000001668. PMID 28514241